CLINICAL TRIAL: NCT01910051
Title: Explorative Assessment of Biomarkers Indicative of Insulin Resistance and Prediabetes in Overweight and Obese Subjects
Brief Title: Explorative Assessment of Biomarkers in Overweight and Obese Subjects
Status: Completed | Type: Observational
Sponsor: Profil Institut für Stoffwechselforschung GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: OBDM-01
Record Dates: First submitted 2013-07-11; First posted 2013-07-29 (Estimated); Last update posted 2021-12-29 (Actual); Status verified 2021-12

CONDITIONS: Prediabetes
MeSH Terms: conditions — Prediabetic State

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Generally healthy: Generally healthy
- Type 2 diabetes mellitus: Type 2 diabetes mellitus

SUMMARY:
The rationale for this trial is to apply a simple and minimally strenuous pre-screening approach prior to performing more extensive trial-specific screening and baseline-characterization activities in the resulting pre-selected population of subjects.

DETAILED DESCRIPTION:
The pre-screening assessments are designed to characterize the metabolic risk profile / prediabetic status in an unselected population of overweight and obese volunteers, aiming to pre-select high risk and prediabetic subjects as a target population who may specifically profit from primary diabetes intervention (prevention) strategies.

ELIGIBILITY:
Inclusion Criteria:

* Obese and overweight subjects
* Considered generally healthy

Exclusion Criteria:

* Clinically significant acute illness within 2 weeks before study procedures

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Generally healthy or Type 2 Diabetes mellitus
Sampling Method: Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2013-09-25 (Actual); Primary Completion 2021-12-23 (Actual); Study Completion 2021-12-23 (Actual)

PRIMARY OUTCOMES:
anthropometric measures and metabolic biomarkers indicative of prediabetes | Day one
  One blood sample taken on day 1 of the study

SECONDARY OUTCOMES:
intra-subject and inter-subject variability of analyzed biomarkers | within one month
  Several circulating markers including the traditionally used fasting serum insulin and fasting plasma glucose as well as an oral glucose tolerance test may serve as indicators of prediabetes. Importantly, these parameters show considerable intra-individual short-term variability. The assessments will therefore be repeated three times within a one month period to determine intra-subject variability of the analyzed parameters under the conditions that apply to the trial site and experimental conditions.

OTHER OUTCOMES:
the correlation between anthropometric data, medical history, and biomarkers with regard to metabolic risk | up to 3 years
  assessment of study data at the end of the study

CONTACTS AND LOCATIONS:
Overall Officials: Leona Plum-Mörschel, MD, Principal Investigator — Profil Institut für Stoffwechselforschung GmbH
Locations (1):
- Profil Institut für Stoffwechselforschung GmbH, Neuss, Germany